CLINICAL TRIAL: NCT06551363
Title: Atopic Dermatitis Cutaneous Discomfort of the Infant Under the Age of One Year : Analysis of Filmed Sequences
Brief Title: Atopic Dermatitis Cutaneous Discomfort of the Infant Under the Age of One Year : Analysis of Filmed Sequences (PRE-PRURINEO)
Acronym: PRE-PRURINEO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0023 - PRE-PRURINEO
Record Dates: First submitted 2019-06-21; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; infant; Etology
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analysis of filmed sequences for the assessment of discomfort in atopic dermatitis in infants under 1year of age

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is a chronic inflammatory and itchy dermatitis particularly common in childhood since it affects about 20% of the pediatric population, with revelation usually around the age of 3-6 months of life. However, there are very few pediatric population data on the prevalence of pruritus and associated discomfort in infants. Although the skin and the nervous system of the infant (<6 months) are competent in the experiment of the pruritus, the acquisition of an intentional motricity allowing the targeted scratching of the affected body areas is done only from the age of 6 months, making it difficult to diagnose the intensity of the AD and assess the potential discomfort caused. Currently, the diagnosis and assessment of pruritus in children is based on a hetero-rating through scales, which are not at all applicable for infants under 6 months of age (population concerned by our study).

The visual scale Numeric Rating Scale, validated in adult population seems to be the one that most accurately assesses the severity of pruritus. In pediatric populations, the use of the Eppendorf Itch Questionnaire and the US version of the Childhood Atopic Dermatitis Impact Scale are recommended. Alternatives to the clinical and subjective rating of the severity of pruritus have been described via actigraphy: thus, a strong statistical correlation has been demonstrated between a nocturnal measurement of wrist motor activity as a reflection of the intensity of pruritus, and the analysis of videos filmed in infra-red. But, again, the technique is not suitable for young infants, because of the absence of voluntary motivated motor skills, and because of less organized sleep / wake cycles.

In order to better manage infants less than 1 year old, the analysis of their behavior in case of atopic dermatitis seems necessary to us to better identify a potential discomfort in these patients.

This is an essential preliminary study that will allow us to better define the judgment criteria necessary for the implementation of an observational study comparing infants with atopic dermatitis to healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 1 year old
* with atopic dermatitis
* No opposition from at least one of the patient's parents

Exclusion Criteria:

* Acute intercurrent pathology
* Severe malformation or genetic abnomalies
* Parent (s) minor (s) or unfit (s) to give their informed consent
* Refusal of patients

Ages: 0 Months to 1 Year | Sex: All
Age Groups: Child
Study Population: Infants with moderate to severe atopic dermatitis less than 1 year old
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Focal sampling and Scan sampling of the behaviors | 6 month
  Frequency of behaviors observed by the method of "focal sampling" and "scan sampling".
  All behavioral responses of the infants will be quantified from the video recordings.

SECONDARY OUTCOMES:
Frequency of behaviors according to the severity of atopic dermatitis | 6 month
  Frequency of focal sampling behaviors according to the severity of atopic dermatitis evaluated using SCORAD score All behavioral responses of the infants will be quantified from the video recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France